CLINICAL TRIAL: NCT06226363
Title: Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetic Characteristics and Initial Efficacy of LNF1901 in Advanced Malignant Tumors
Brief Title: Phase I Study of LNF1901 in Advanced Malignant Tumors
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shandong New Time Pharmaceutical Co., LTD (Industry)
Collaborators: Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NTP-LNF1901-001
Record Dates: First submitted 2024-01-17; First posted 2024-01-26 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Advanced Malignant Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LNF1901 monotherapy (Experimental)
  Interventions: Drug: LNF1901 Monoclonal Antibody Injection

INTERVENTIONS:
Drug: LNF1901 Monoclonal Antibody Injection — LNF1901，7 dose groups:0.003mg/kg、0.03mg/kg、0.1mg/kg、0.3mg/kg、1mg/kg、2mg/kg、3mg/kg，IV, infusion time 60min±10min, Q3W, until disease progression or other reasons to stop treatment, the longest administration to 2 years, whichever occurs first.

SUMMARY:
This is a multicenter, open, phase I dose-escalation and dose-expansion study to evaluate the safety, tolerability, initial antitumor efficacy, PK and immunogenic characteristics of LNF1901 in patients with advanced malignancies.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18 years of age;
2. Patients with advanced malignant tumors who have been confirmed histologically or cytologically and have failed to receive standard therapy, or cannot tolerate standard therapy, or cannot receive standard therapy for other reasons;
3. Participants enrolled in the dose expansion phase had at least one measurable lesion; (4) Those who adopted the United States Eastern Oncology Consortium (ECOG) physical status score of 0~1;

5) The researchers judged that the expected life of the subjects was ≥3 months; 6) The function of vital organs meets the following requirements (drugs with blood components and cytokines are not allowed to be used within 14 days before the first administration) : Blood routine: Absolute neutrophil count (ANC) ≥1.5×109/L; Platelet count ≥80×109/L; Hemoglobin (Hb) ≥90g/L; Liver function: aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤2.5×ULN, serum total bilirubin (TBIL) ≤1.5×ULN; If liver metastasis exists, AST and ALT≤5×ULN, TBIL≤1.5×ULN; Renal function: serum creatinine (Cr) ≤1.5×ULN or creatinine clearance ≥50mL/min (Cr > 1.5×ULN); Coagulation function: International Normalized ratio (INR) ≤1.5×ULN and activated partial thromboplastin time (APTT) ≤1.5×ULN; Thyroid function: Thyroid stimulating hormone (TSH) within the normal range or free triiodothyronine (FT3), free thyroxine (FT4) normal or abnormal without clinical significance; 7) Subjects voluntarily participate in the study and sign the informed consent after receiving full informed consent.

Exclusion Criteria:

1. Those who have previously received antibody treatment with any tumor necrosis factor receptor (TNFR) superfamily agonists, such as CD40, OX40, CD137, CD27, CD357, etc.;
2. Those who have received anti-tumor therapy 4 weeks before the first administration or within 5 half-lives of the drug (whichever is shorter);
3. Chronic systemic glucocorticoid therapy within 2 weeks prior to initial administration (daily dose equivalent to prednisone > 10mg of systemic corticosteroids) or any other form of immunosuppressive therapy;
4. The toxicity of previous anti-tumor therapy has not returned to CTCAE5.0 version of the definition ≤ Class 1 (except hair loss);
5. A history of cancer within the past 5 years, except for locally curable cancers (radical melanoma, basal or squamous cell carcinoma, carcinoma in situ of the bladder or cervix);
6. Patients with primary central nervous system (CNS) malignancies, CNS metastases after local treatment failure, and cancerous meningitis; Patients with asymptomatic brain metastases or stable neurological symptoms without steroid hormones or other BMS for ≥4 weeks could be enrolled.
7. Patients with a history of organ transplantation or allogeneic bone marrow transplantation or who have received autologous stem cell transplantation within 3 months before the first administration of the drug;
8. Those who have undergone major surgery or have not recovered from surgery within 4 weeks prior to the first dosing (except for diagnostic surgery);
9. Physical examination or laboratory examination, any of the following conditions:

   Hepatitis B: HBsAg positive and/or HBcAb positive with HBV-DNA titers positive or higher than the upper limit of normal (excluded if only the lower limit of detection is present); Hepatitis C: HCV antibody positive and HCV-RNA positive or greater than the upper limit of normal; Human immunodeficiency virus (Anti-HIV) positive; active treponema pallidum infection;
10. Uncontrolled or severe cardiovascular disease, such as New York Heart Association (NYHA) Class II or above congestive heart failure, unstable angina, myocardial infarction and other cardiovascular disease, poorly controlled arrhythmias, within 6 months before the first administration of the drug. Difficult to control hypertension (systolic blood pressure ≥160mmHg and/or diastolic blood pressure ≥100mmHg after adequate treatment);
11. Patients with a history of the following, including but not limited to active autoimmune diseases, active infections (such as active tuberculosis), severe mental illness, and severe endocrine disorders;
12. Patients who have been treated with any other investigational drug/device within 4 weeks prior to initial administration;
13. Have a history of drug abuse or alcoholism within 6 months before the first dose;
14. Have a history of severe allergy, and known subjects are previously allergic to macromolecular protein preparations/monoclonal antibodies and to any investigational drug components;
15. Those who received live or attenuated vaccine within 4 weeks before the first dose or planned to receive live or attenuated vaccine during the study period;
16. Pregnant or lactating women, female subjects of childbearing age, or male subjects whose partners are women of childbearing age who do not consent to the use of medically approved effective contraceptive methods (such as Iuds or condoms) during the study period and within 6 months after the last study drug treatment;
17. Those who were judged not suitable for inclusion by the researchers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities | Up to 21 days following first dose of APX005M
  DLTs will include Grade 4 neutropenia, anemia, thrombocytopenia, Grade 4 cytokine release syndrome and other Grade 3 non-hematological toxicity etc
Incidence of adverse events | Through up to approximately 30 days following last dose of LNF1901
  Incidence and severity of AEs and specific laboratory abnormalities graded according to NCI-CTCAE, v5.0